CLINICAL TRIAL: NCT06311721
Title: A Randomized, Double-Blind Study to Compare Efficacy, Pharmacokinetics, Safety, and Immunogenicity Between ABP 234 and Keytruda® (Pembrolizumab) in Subjects With Advanced or Metastatic Non-squamous Non-Small Cell Lung Cancer
Brief Title: A Study to Compare ABP 234 and Keytruda® (Pembrolizumab) in Participants With Advanced or Metastatic Non-squamous Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20210033; 2023-508336-57 (EudraCT Number); 2024-514304-14-00 (Other: EUCTR)
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Advanced or Metastatic Non-squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ABP 234 (Experimental): Part 1: Participants will receive ABP 234 followed by pemetrexed administered with platinum-based chemotherapy (cisplatin or carboplatin). Part 2: Participants will receive ABP 234 followed by pemetrexed.
  Interventions: Drug: ABP 234
- Pembrolizumab (US) (Experimental): Part 1: Participants will receive FDA-licensed pembrolizumab followed by pemetrexed administered with platinum-based chemotherapy (cisplatin or carboplatin). Part 2: Participants will receive FDA-licensed pembrolizumab followed by pemetrexed.
  Interventions: Drug: Pembrolizumab (US)
- Pembrolizumab (EU) (Experimental): Part 1: Participants will receive EU-approved pembrolizumab followed by pemetrexed administered with platinum-based chemotherapy (cisplatin or carboplatin). Part 2: Participants will receive EU-approved pembrolizumab followed by pemetrexed.
  Interventions: Drug: Pembrolizumab (EU)

INTERVENTIONS:
Drug: ABP 234 — Intravenous administration
  Arms: ABP 234
Drug: Pembrolizumab (US) — Intravenous administration
  Other Names: Keytruda®
  Arms: Pembrolizumab (US)
Drug: Pembrolizumab (EU) — Intravenous administration
  Other Names: Keytruda®
  Arms: Pembrolizumab (EU)

SUMMARY:
The primary objective of this study is to compare the efficacy of ABP 234 with the pembrolizumab reference product (Keytruda®).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Histologically or cytologically confirmed stage IV non-squamous Non-Small Cell Lung Cancer (NSCLC).
3. Participant has no prior systemic treatment for advanced disease.
4. Measurable disease according to RECIST v1.1.
5. Tumor tissue from the resected site of disease must be available for biomarker analyses in order to be randomized.
6. Eastern Cooperative Oncology Group performance status score 0 or 1.
7. Epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), and c-ros oncogene 1, receptor tyrosine kinase of the insulin receptor family (ROS-1) negative
8. Have a life expectancy of at least 3 months.

Exclusion Criteria:

1. Small cell lung cancer (SCLC) or mixed SCLC/NSCLC histology or squamous cell carcinoma.
2. Participant has active central nervous system metastases not previously treated.
3. Participant has active or known immune-mediated disorders.
4. Participant has received prior systemic cytotoxic chemotherapy, immunotherapy (including PD-1/PD-L1), anti-neoplastic biological therapy, or targeted therapy for advanced/metastatic disease.
5. Known hypersensitivity to monoclonal antibodies or to any of the excipients of the study drug, or to any component of cisplatin, carboplatin, or pemetrexed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2028-02-14 (Estimated); Study Completion 2028-05-29 (Estimated)

PRIMARY OUTCOMES:
Objective response (OR) | Week 49
  OR defined as an overall response of confirmed complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Area under the serum concentration-time curve (AUC) from time 0 to 21 days (AUC21d) of ABP 234 | 21 days
AUC at steady state between Week 16 and Week 19 (AUCtau_ss) of ABP 234 | Week 16 through Week 19

SECONDARY OUTCOMES:
OR | Week 13
OR | Week 31
Duration of response (DOR) | Up to 2.5 years
Progression-free survival (PFS) | Up to 2.5 years
Overall survival (OS) | Up to 2.5 years
Maximum observed serum concentration following the first dose (Cmax_dose1) of ABP 234 | Day 1 up to Week 107
Cmax_dose1 of pembrolizumab (US) | Day 1 up to Week 107
Cmax_dose1 of pembrolizumab (EU) | Day 1 up to Week 107
Time to maximum concentration following the first dose (tmax_dose1) of ABP 234 | Day 1 up to Week 107
Tmax_dose1 of pembrolizumab (US) | Day 1 up to Week 107
Tmax_dose1 of pembrolizumab (EU) | Day 1 up to Week 107
Maximum observed serum concentration (Cmax) at steady state (Cmax_ss) of ABP 234 | Week 16 through Week 19
Cmax_ss of pembrolizumab (US) | Week 16 through Week 19
Cmax_ss of of pembrolizumab (EU) | Week 16 through Week 19
Time to maximum concentration at steady state (tmax_ss) of ABP 234 | Week 16 through Week 19
Tmax_ss of pembrolizumab (US) | Week 16 through Week 19
Tmax_ss of pembrolizumab (EU) | Week 16 through Week 19
Trough serum concentrations at pre-dose of week 4 (Ctrough_w4) of ABP 234 | Week 4
Ctrough_w4 of pembrolizumab (US) | Week 4
Ctrough_w4 of pembrolizumab (EU) | Week 4
Trough serum concentrations at steady state (Ctrough_ss) at pre-dose of ABP 234 | Week 16 through Week 19
Ctrough_ss at pre-dose of pembrolizumab (US) | Week 16 through Week 19
Ctrough_ss at pre-dose of pembrolizumab (EU) | Week 16 through Week 19
AUC21d of pembrolizumab (US) | 21 days
AUC21d of pembrolizumab (EU) | 21 days
AUCtau_ss of pembrolizumab (US) | Week 16 through Week 19
AUCtau_ss pembrolizumab (EU) | Week 16 through Week 19
Number of participants who experience a Treatment-emergent adverse event | Up to 2.5 years
Number of participants who experience a Treatment-emergent serious adverse event | Up to 2.5 years
Number of participants who experience a Treatment-emergent adverse event of interest | Up to 2.5 years
Number of participants who experience anti-drug antibodies (ADA) | Up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (219):
- United States (15):
  - Precision NextGen Oncology and Research Center, Beverly Hills, California
  - TOI Clinical Research, Cerritos, California
  - Cancer and Blood Specialty Clinic (CBSC), Los Alamitos, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - PIH Health Hospital, Whittier, California
  - Millennium Oncology - Hollywood, Hollywood, Florida
  - BRCR Medical Center Inc., Tamarac, Florida
  - Accellacare Duly, Plainfield, Illinois
  - Accellacare of McFarland, Ames, Iowa
  - Detroit Clinical Research Center, PC, Farmington Hills, Michigan
  - North Shore Hematology-Oncology Associates P.C. d/b/a New York Cancer & Blood Specialists, Shirley, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - Millennium Research and Clinical Development, LLC, Houston, Texas
  - Texas Oncology, P.A, San Antonio, Texas
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Wytheville, Virginia
- Argentina (6):
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Buenos Aires
  - Centro de Investigacion Pergamino SA, Pergamino, Buenos Aires
  - Fundacion ARS Medica, San Salvador de Jujuy, Jujuy Province
  - Sanatorio Britanico De Rosario, Rosario, Santa Fe Province
  - Hospital Provincial del Centenario, Rosario, Santa Fe Province
  - IONC - Instituto Oncologico de Cordoba, Córdoba
- Austria (2):
  - Klinikum Klagenfurt am Woerthersee, Klagenfurt
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
- Brazil (36):
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - OC Oncoclinicas Oncovida, Brasília, Destrito Federal
  - Centro de Pesquisas Clinicas em Oncologia (CPCO)/HECI, Cachoeiro de Itapemirim, Espírito Santo
  - Associacao Feminina de Educacao e Combate ao Cancer(AFECC) - Hospital Santa Rita, Vitória, Espírito Santo
  - Hospital Santa Izabel, Santa Casa de Misericordia da Bahia, Salvador, Estado de Bahia
  - Cetus Oncologia S.A. Unidade Belo Horizonte, Belo Horizonte, Minas Gerais
  - Nucleo de Ensino Pesquisa e Inovacao Mario Penna, Belo Horizonte, Minas Gerais
  - Fundacao Sao Francisco Xavier - Hospital Marcio Cunha (HMC) - Unidade I, Ipatinga, Minas Gerais
  - Liga Paranaense de Combate ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - Instituto de Cancer de Londrina - Hospital do Cancer de Londrina - HCL, Londrina, Paraná
  - Liga Contra o Cancer, Natal, Rio Grande do Norte
  - Hospital Tacchini, Bento Gonçalves, Rio Grande do Sul
  - Oncosite Centro De Pesquisa Clinica Em Oncologia, Ijuí, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital da Cidade de Passo Fundo - HCPF, Passo Fundo, Rio Grande do Sul
  - Unidade de Pesquisa Clinica em Oncologia Ltda (UPCO) (Clinica Lacks), Pelotas, Rio Grande do Sul
  - Centro de Pesquisa em Oncologia - Hospital Sao Lucas da PUC Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Associacao dos Functionarios Publicos do Estado do Rio Grande do Sul - Hospital Ernesto Dornelles (H, Porto Alegre Rio Grande Do Sul, Rio Grande do Sul
  - Centro de Oncologia de Santa Catarina Ltda / Supera Oncologia, Chapecó, Santa Catarina
  - CEPEN Centro de Pesquisa e Ensino em Saude de Santa Catarina, Florianópolis, Santa Catarina
  - Instituto Joinvillense de Hematologia e Oncologia SS Ltda - Clinica de Hematologia e Oncologia, Joinville, Santa Catarina
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Centro de Pesquisa Sao Lucas, Campinas, São Paulo
  - Centro Oncologico Mogi das Cruzes, Mogi das Cruzes, São Paulo
  - Instituto Ribeiraopretano de Combate ao Cancer (IRPCc) - IRPCC, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC - Centro de Estudos e Pesqulsas de Hematologia e Oncologia, Santo André, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto - Hospital de Base de Sao Jose do R, São José do Rio Preto, São Paulo
  - Hospital Nossa Senhora das Gracas, Canoas
  - CIONC - Centro Integrado de Oncologia de Curitiba, Curitiba
  - Centro Integrado de Pesquisa em Oncologia - Hospital Nossa Senhora da Conceio, Porto Alegre
  - Instituto Nacional de Cancer (INCA), Rio de Janeiro
  - Instituto Americas - Ensino, Pesquisa e Inovacao, Rio de Janeiro
  - Oncoclinicas Rio de Janeiro S.A (Centro de Tratamento de Tumores Botafogo), Rio de Janeiro - RJ
  - Instituto D'Or de Pesquisa e Ensino - Hospital Sao Rafael, Salvador
  - Hospital Alemao Oswaldo Cruz (HAOC), São Paulo
  - Instituto Brasileiro de Controle do Cancer - IBCC Oncologia, São Paulo
- Bulgaria (3):
  - University Multi-Profile Hospital for Active Treatment (UMHAT) St. Ivan Rilski, Sofia, Sofia-Grad
  - MHAT Dobrich AD, Dobrich
  - University Multiprofile Hospital for Active Treatment Sofiamed, Sofia
- Chile (7):
  - Oncocentro, Viña del Mar, Región de Valparaíso
  - Centro de Investigaciones Clinicas Vina del Mar Ltda., Viña del Mar, Región de Valparaíso
  - CDIEM - Centro de Investigacion y Especialidades Medicas, Providencia, Santiago Metropolitan
  - Centro de Oncologa de Precisin, Region Metropolitana, Santiago Metropolitan
  - Clinica Santa Maria, Santiago, Santiago Metropolitan
  - K2 Oncology, Santiago
  - Icegclinic Research and Care, Santiago
- France (8):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Saint - Andre, Bordeaux
  - Centre Hospitalier Universitaire (CHU) De Limoges Hopital Dupuytren, Limoges
  - Hopital Europeen Marseille, Marseille
  - Clinique Clementville-Gcs Centre De Cancerologie Du Grand Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nimes (CHU) - Hopital Universitaire Caremeau, Nîmes
  - Centre Hospitalier Intercommunal Toulon La Seyne Sur Mer (C.H.I.T.S) - Hospital Font-Pre, Toulon
  - Clinique Teissier, Valenciennes
  - Hopital Robert Schuman, Vantoux
- Georgia (6):
  - High Technology Hospital Medcenter LTD, Batumi
  - Israel-Georgian Medical Research Clinic Healthycore, Tbilisi
  - LLC Todua Clinic, Tbilisi
  - TIM -Tbilisi Institute of Medicine, Tbilisi
  - New Hospitals, Tbilisi
  - Medulla - Clinics And Medical Centers, Tbilisi
- Germany (4):
  - Evang. Kliniken Essen Mitte GmbH, Essen
  - Studienzentrum Aschaffenburg, HÃ¶sbach
  - Haematologie, Onkologie und Palliativmedizin, Tagesklinik Landshut, Landshut
  - FEK - Friedrich-Ebert-Krankenhaus Neumuenster GmbH, Neumünster
- Italy (8):
  - Azienda Ospedaliero - Universitaria di Ferrara, Cona
  - Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Fondazione Irccs Ca' Granda Ospedale Maggiore Policlinico Di Milano, Milan
  - UOC Oncoematologia AOU Luigi Vanvitelli, Naples
  - ASL Napoli 1 Centro-Ospedale del Mare, Napoli
  - AUSL Della Romagna - Ospedale S.Maria delle Croci, Ravenna
  - S.C. Oncologia Medica-Presidio Ospedaliero Sondrio, Sondrio
  - Azienda Ospedaliera Santa Maria Terni, Terni
- Japan (21):
  - Japan Community Healthcare Organization Chukyo Hospital, Nagoya, Aichi-ken
  - Funabashi Municipal Medical Center, Funabashi-shi, Chiba
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Aso Iizuka Hospital, Iizuka-shi, Fukuoka
  - Japanese Red Cross Maebashi Hospital, Maebashi, Gunma
  - Chugoku Central Hospital, Fukuyama, Hiroshima
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Asahikawa Medical University Hospital, Asahikawa, Hokkaido, Japan
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki, Hyōgo
  - Nippon Medical School Musashikosugi Hospital, Kawasaki-shi, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Yokosuka Kyosai Hospital, Yokosuka, Kanagawa
  - Social Welfare Organization Imperial Gift Foundation, Inc. Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Osaki Citizen Hospital, Ōsaki, Miyagi
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki, Miyazaki
  - Shinshu University Hospital, Matsumoto, Nagano
  - NHO Kinki Chuo Chest Medical Center, Sakai, Osaka Japan
  - Kawaguchi Municipal Medical Center, Kawaguchi-shi, Saitama
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Hamamatsu Medical Center, Hamamatsu, Shizuoka, Japan
  - Ome Medical Center, Ome-shi, Tokyo
- Malaysia (5):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Raja Perempuan Zainab II Hospital, Kota Bharu, Kelantan
  - Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur
  - Sarawak General Hospital, Kuching, Sarawak
  - University of Malaya Medical Centre, Kuala Lumpur
- Peru (7):
  - Hospital III Goyeneche, Cercado, Arequipa
  - Instituto Nacional De Enfermedades Neoplasicas, Surquillo, Lima, Peru
  - Hospital IV - Alberto Sabogal Sologuren Red Asistencial Sabogal, Bellavista, Provincia Constitucional del Callao
  - Centro Medico Monte Carmelo, Arequipa
  - Clinic Vallesur Arequipa, Arequipa
  - Hospital de Apoyo Maria Auxiliadora, Lima
  - Clnica San Antonio, Trujillo
- Philippines (11):
  - Cebu Doctors University Hospital, Cebu City, Cebu
  - Chong Hua Hospital, Cebu City, Cebu
  - Perpetual Succour Hospital, Cebu City, Central Visayas
  - Davao Doctors Hospital, Davao City, Davao Del Sur
  - West Visayas State University Medical Center, Iloilo City, Iloilo
  - Asian Hospital And Medical Center, Muntinlupa, National Capital Region
  - Veterans Memorial Medical Center, Quezon City, National Capital Region
  - St. Lukes Medical Center, Quezon City, NCR
  - Riverside Medical Center Inc, Bacolod City, Negros Occidental
  - St. Paul's Hospital of Iloilo, Inc., Iloilo City, Western Visayas
  - Philippine General Hospital, Manila
- Poland (7):
  - Centrum Onkologii im. Prof. F. Lukaszczyka w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin, Lublin Voivodeship
  - Warminsko Mazurskie Centrum Chorob Pluc w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
  - Instytut MSF Sp. z o.o., Lodz
  - NZOZ Neuromed M. i M. Nastaj Sp.P, Lublin
  - Med-Polonia Sp. z o.o., Poznan
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku Sp. z o.o., Słupsk
- Serbia (3):
  - Clincial Centre of Serbia, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - University Clinical Centre of Kragujevac, Kragujevac
- South Africa (5):
  - GVI Oncology, Langenhoven Drive Oncology Centre, Port Elizabeth, Eastern Cape
  - University of Pretoria and Steve Biko Academic Hospital Complex, Pretoria, Gauteng
  - Life Wilgers Hospital Wilgers Oncology Centre, Pretoria, Gauteng
  - Dr W M Szpak Inc - Rainbow Oncology, Athlone Park, KwaZulu-Natal
  - Abraham Oncology, Richards Bay, KwaZulu-Natal
- South Korea (9):
  - The Catholic University Of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Jeonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (15):
  - Hospital General Universitario de Elche, Alicante
  - UOMI Cancer Center-Clinica Tres Torres, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Complejo Hospitalario de Jaen (University Hospital Ciudad De Jaen), Jaén
  - Hospital Universitario San Francisco de Asis, Madrid
  - Hospital Unifersitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Fundacion Alcorcon, Madrid
  - Hospital De Mataro, Mataró
  - Hospital Quironsalud Malaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Nuestra Senora De Valme, Seville
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulev, Valencia
  - Hospital Quironsalud Valencia, Valencia
- Taiwan (11):
  - Tri-Service General Hospital, Neihu, Taipei
  - National Taiwan University Hospital (NTUH), Taipei, Zhongzheng Dist
  - Dalin Tzu chi General Hospital - Buddhist Tzu chi Medical Foundation, Chiayi City
  - National Taiwan University Hospital Yun-Lin Branch, Douliu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation Kaohsiung Chang Gung Memorial Hospital, Kaohsiung County
  - Taipei Medical University (TMU) - Shuang Ho Hospital (SHH), New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- Thailand (8):
  - Mahidol University - Siriraj Hospital - Siriraj Clinical Research Center (SICRC), Bangkoknoi, Bangkok
  - Chiangrai Prachanukroh Hospital, Muang, Changwat Chiang Rai
  - Naresuan University Hospital, Muang, Changwat Phitsanulok
  - Prince Of Songkla Hospital, Prince Of Songkhla University, Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai University, Muang, Chiang Mai
  - Chulabhorn Hospital, Talat Bang Khen, Lak Si
  - Faculty of Medicine Vajira Hospital, Navamindradhiraj University, Bangkok
  - King Chulalongkorn Memorial Hospital, Chulalongkom University, Bangkok
- Turkey (Türkiye) (21):
  - Adana Ortadogu Hospital, Seyhan, Adana
  - Gulhane Training and Research Hospital, Keçiören, Ankara
  - Gazi University Faculty of Medicine, Yenimahalle, Ankara
  - Trakya University Faculty of Medicine, İskender, Edirne
  - Ondokuz Mayis University Health Practice and Research Hospital, Atakum, Samsun
  - Medical Park Seyhan Hospital, Adana
  - Adana City Training and Research Hospital, Adana
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, Ankara
  - Memorial Ankara Hospital, Ankara
  - Liv Hospital Ankara, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Uludag University Medical Faculty, Bursa
  - Medical Point Gaziantep Hospital, Gaziantep
  - Bezmialem Foundation University Medical Faculty, Istanbul
  - Yeditepe University Kosuyolu Hospital, Istanbul
  - Istanbul Medeniyet University Medical Faculty, Istanbul
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Sakarya Universitesi Tip Fakultesi, Sakarya
  - Namik Kemal Universitesi Hastanesi, Tekirdağ
- Nottingham University Hospitals NHS Trust - Nottingham City Hospital, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com